CLINICAL TRIAL: NCT02792140
Title: The Impact of the Opiate Antagonist Naltrexone on the Emotional Valence of Dreams
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015DR2186
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Neuroscience of Dreaming, Healthy
Keywords: Psychology; Dreams
MeSH Terms: interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Baseline (No Intervention): reporting of dreams
- Naltrexone (Experimental): daily administration of 50mg Naltrexone, reporting of dreams
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): daily administration of Placebo, reporting of dreams
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naltrexone — one week
  Other Names: Naltrexin
  Arms: Naltrexone
Other: Placebo — one week
  Other Names: Placebo Pills
  Arms: Placebo

SUMMARY:
In this study, the investigators pose the question which influence the opioid circuit has on positive valent situations in dreams.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthiness
* Good capacity of remembering dreams
* No opiate consumption

Exclusion Criteria:

* Simultaneous participation in other studies
* Addictive disorder
* Abnormal liver function
* Abnormal kidney function
* Hypersensitivity to active ingredient or pharmaceutical additives
* Hereditary galactose intolerance
* Lactase deficiency
* Glucose-galactose malabsorption
* Intake of opioid medication

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
VAS-difference concerning the emotional valence of dreams | 7 days per condition (Naltrexone, Placebo), intermitted by 14 days of washout
  Difference between the mean values of emotional valence of dreams reported in the conditions (Naltrexone, Placebo), as captured in VAS [visual analog scales] for every dream

SECONDARY OUTCOMES:
Semiquantitative score of emotional valence of dreams | 7 days per condition (Baseline, Naltrexone, Placebo), intermitted by 14 days of washout
  Based on computational linguistic analysis of the dreams
Qualitative score of emotional valence of dreams | 7 days per condition (Baseline, Naltrexone, Placebo), intermitted by 14 days of washout
  Based on lexical coding of the dreams

CONTACTS AND LOCATIONS:
Overall Officials: Fred Mast, Prof. Dr. phil., Study Director — Head of Cognitive Psychology, Perception and Research Methods, Dean Human Sciences Faculty, Ordinarius, University of Bern; Claudio L. Bassetti, Prof. Dr. med., Principal Investigator — Chairman and Head, Department of Neurology Inselspital, Bern University Hospital
Locations (1):
- University of Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided